CLINICAL TRIAL: NCT03914482
Title: Feasibility Study to Estimate Fat Concentration of Liver in Adults Through RF Imaging
Brief Title: Fatty Liver Imaging Project ( FLIP ) Patient Pilot Study
Acronym: FLIP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The qualified and Principal Investigator has moved institutes. We are in the process for finding a replacement.
Sponsor: Aaron Fenster (Other)
Collaborators: Endra Lifesciences (Industry)
Responsible Party: Sponsor-Investigator, Aaron Fenster, Scientist, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6186
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients at risk of FLD (Other): Patients who choose to participate in the study that meet the inclusion criteria
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — The device will acquire thermoacoustic data while the ultrasound probe acquires ultrasound images, and an MR of the liver is acquired as a comparative modality
  Other Names: Liver Imaging

SUMMARY:
This study is being done to test the FLIP device, a novel device developed and manufactured by Endra Life Sciences, located in Ann Arbor, Michigan. The purpose of the device is to measure the fat content of liver tissue to assist in the diagnosis of fatty liver disease. This feasibility study will involve 50 patients having their liver imaged by traditional ultrasound and MRI methods as well as using the FLIP device. The data obtained by the FLIP will be compared with the data obtained by ultrasound and MRI in order to determine the effectiveness of the device. This is a preliminary study to see if the investigational device could eventually be used to image the liver alongside traditional ultrasound for discerning fat concentration.

DETAILED DESCRIPTION:
It has been demonstrated that thermoacoustic imaging can be used to identify water and fat concentrations [Bauer, 2012]. In addition, the group led by Dr. Kruger have demonstrated that conventional computed tomography shows similar features to thermoacoustic imaging in small animal studies [Kruger, 2003]. These concepts have led Endra Life Sciences to develop the FLIP device with the purpose of imaging fat concentration in liver tissue with indications for fatty liver disease. Non-alcoholic fatty liver disease (NAFLD) was first reported in 1980 by pathologists at the Mayo clinic in obese, or overweight, patients with no history of alcohol abuse. This represented the first time that fatty livers were observed with no history of alcohol abuse. Since that first report of NAFLD, increased rates of obesity and general increased caloric intake has dramatically increased rates of fatty liver disease. Estimates of NAFLD range from 25 - 40% of the adult population globally. NAFLD is a multi-system disease. Fatty liver disease is highly correlated with obesity and alcohol abuse, and is an important biomarker of insulin resistance and metabolic disease. Endra's technology offers a non-invasive, cost effective point of care solution to monitoring liver fat content that will be enormously helpful in surveilling patients with metabolic disease, insulin resistance, and those at risk for later stage liver disease. This study will provide additional information that will guide the further development of the FLIP device with the end goal of commercializing the product. Fibroscan is a device that is currently on the market that is also indicated for fatty liver disease. Fibroscan is a shear wave elastography device that measures the stiffness of liver tissue by mechanically deforming tissue (by utilizing a plunger that vibrates the surface of the skin) and measures the resulting shear wave speed within the liver by ultrasound. The shear wave speed is related to the mechanical stiffness of the tissue. Fibroscan aims to assess the progression of infiltration of collagen into normal liver tissue that results in scarring, characteristic of fibrotic liver disease. Liver fibrosis progresses from fatty liver disease, not all fatty liver disease patients develop fibrotic liver disease. The Fibroscan device has an optional software module that attempts to quantify the attenuation of the shear wave as it travels away from the plane of deformation. Fibroscan refers to this measurement as CAP (Calculated Attenuation Parameter). The attenuation of the shear wave is thought to be related to the degree of liver steatosis (fat content).

To date, the technique has demonstrated poor sensitivity, and is poorly correlated with quantitative MRI measures of liver fat. Furthermore, CAP measurements in obese patients are difficult to obtain and unreliable. Endra's technology aims to provide much more sensitive measurements of liver fat content at the point of care. The Endra device has the potential to quantify fat content as low as 5% (by volume). The system is interoperable with ultrasound and leverages B-mode ultrasound imaging to guide measurement location. Compared to Fibroscan's CAP, Endra's fatty liver measures are expected to be much more sensitive and reproducible based on anatomical guidance by ultrasound imaging.

A healthy volunteer study was conducted to test the overall feasibility of the device in use in humans. The median liver fat percentage was in the normal range, less than six percent, which helped gauge the accuracy of using the device in detecting low levels of liver fat. In addition, the operator was able to optimize the use of the device on human scanning. Of the 25 study subject datasets analyzed, only 4 subjects had above normal liver fat by MRI fat fraction (normal is < 6% fat fraction). All 4 study subjects with >6% liver fat fraction, fell into 'mild liver fat' grade that spans 6% - 26% fat fraction, with the maximum value of 22%.

Using all 25 study subject datasets the TAEUS investigational device measurement has an R^2 correlation value of 0.61 with MRI measurements of fat fraction. This is particularly interesting as BMI and abdominal fat thickness were found to have R^2 correlation values with MRI measures of liver fat of 0.19 and 0.31, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients which have had at least 1 appointment with a clinician for liver function, diabetes, or obesity in the past year.
* Must be over the age of 18.
* Mild (6-26%), moderate (26-37%), or high (>37%) level of fat in the liver that is estimated by ultrasound imaging.
* Must be proficient in English (reading/writing).

Exclusion Criteria:

* Any metal or electronic implants including but not limited to pacemakers, metal clips, hips.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Fat concentration estimate | Up to 1 month following data collection
  The purpose of the device is to measure the fat content of liver tissue to assist in the diagnosis of fatty liver disease

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided